CLINICAL TRIAL: NCT03776422
Title: Homeless Youth Study - Stepping Stone 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Illinois Department of Human Services (Unknown); Sparrow Mobile (Unknown)
Responsible Party: Principal Investigator, Alyson Zalta, Assistant Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17072403
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Mental Health Issue (E.G., Depression, Psychosis, Personality Disorder, Substance Abuse)
MeSH Terms: conditions — Depression; Psychotic Disorders; Personality Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile self-help intervention (Experimental): This study uses automated self-help interventions designed as a kit of smartphone tools.
  Interventions: Behavioral: Mobile self-help intervention

INTERVENTIONS:
Behavioral: Mobile self-help intervention — Participants receive several apps on their phone including IntelliCare apps, which are based on principles of cognitive-behavioral therapy. Participants also receive the Pocket Helper app, which has been designed for this study. The tools within the Pocket Helper app include a crisis text line that is available 24/7, the Illinois Warm Line which is available Monday through Friday from 8am to 5pm, directions to call 911 in the case of an emergency, the Koko web app that provides crowdsourced emotional support, brief cognitive-behavioral interventions, daily tips, and daily surveys. Phones will also include the StreetLight Chicago app, which provides homeless individuals with up-to-date information on shelters, health clinics, emergency contacts, mental health services, and more.

SUMMARY:
Housing instability is both a cause and consequence of mental health problems. As such youth experiencing housing instability (e.g., homeless or marginally housed) have higher rates of mental health problems.Because of their circumstances, these youth also face significant barriers to mental health care and are therefore less likely to receive the treatment that they need. Mobile technology may offer a novel platform for increasing access to mental health care in this population. The primary goals of this pilot study are to (1) establish the feasibility and acceptability of delivering automated mental health interventions via smartphone technology, (2) examine the extent to which automated mental health interventions delivered via mobile technology improve mental health in homeless, marginally-housed, and exiting foster youth.

ELIGIBILITY:
Inclusion Criteria:

* 16-25 years
* English-speaking
* Youth must meet one of the following risk criteria

  * Experiencing housing instability as defined by:

    * lacking a fixed, regular, and adequate nighttime residence OR whose primary nighttime residence is a shelter, institution, or a "public or private place not designed for, or ordinarily used as, a regular sleeping accommodation for human beings"
    * sharing the housing of other persons due to loss of housing [or] economic hardship.
    * frequent moves, poor housing quality (e.g., living in severely overcrowded housing).
  * Imminently leaving the foster care system
* Willingness and ability to comply with requirements of the study protocol

Exclusion Criteria:

* Inability to understand study procedures and participate in the informed consent process.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Program adherence | Baseline to Endpoint (6 months)
  Program adherence will be assessed based on usage data determining how often participants utilized the study applications, and how often they completed daily surveys and rated daily tips.
Program satisfaction | Midpoint (3 months) and Endpoint (6 months)
  Program satisfaction will be assessed using a self-report questionnaire that participants will be asked to complete at the midpoint and endpoint of the study. Participants will be asked to report the extent to which they benefited from the study, how helpful the mobile applications were, and if they would recommend the study to others. These responses are recorded on 5-point likert type scales with higher ratings indicating higher satisfaction.

SECONDARY OUTCOMES:
Anxiety symptoms | Baseline (0 months), Midpoint (3 months), Endpoint (6 months)
  Anxiety symptoms will be assessed using the adaptive PROMIS Bank v1.0 for anxiety.
Depression symptoms | Baseline (0 months), Midpoint (3 months), Endpoint (6 months)
  Depression symptoms will be assessed using the adaptive PROMIS Bank v1.0 for depression.
Alcohol use | Baseline (0 months), Midpoint (3 months), Endpoint (6 months)
  Alcohol use will be assessed using the Alcohol Use Disorders Identification Test (AUDIT-C).
Cannabis use | Baseline (0 months), Midpoint (3 months), Endpoint (6 months)
  Cannabis use will be assessed using the Cannabis Use Disorder Identification Test - Revised (CUDIT-R).
Risky sexual behavior | Baseline (0 months), Midpoint (3 months), Endpoint (6 months)
  Risky sexual behaviors will be assessed using the sexual behavior items from the Centers for Disease Control and Prevention's Youth Risk Behavior Survey (2011).
PTSD symptoms | Baseline (0 months), Midpoint (3 months), Endpoint (6 months)
  PTSD symptoms will be assessed using the The Primary Care PTSD Screen for DSM-5 (PC-PTSD-5).
Satisfaction with life: Satisfaction with Life Scale (SWLS) | Baseline (0 months), Midpoint (3 months), Endpoint (6 months)
  General satisfaction with life will be assessed using the Satisfaction with Life Scale (SWLS). This measure is 5 items, with each item rated on a scale from 1-7. All 5 items are summed to achieve a total score of 5-35. Higher scores indicate higher satisfaction with one's life circumstances.
Psychosocial flourishing | Baseline (0 months), Midpoint (3 months), Endpoint (6 months)
  Psychological resources and strengths will be assessed using the Flourishing Scale (FS). This measure is 8 items, with each item rated on a scale from 1-7. All 8 items are summed to achieve a total score of 8-56. Higher scores indicate that an individual has more psychological resources and strengths.

CONTACTS AND LOCATIONS:
Overall Officials: Alyson K Zalta, PhD, Study Director — University of California, Irvine
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Straka K, Blacketer AR, Martinez RL, Glover A, Winiarski DA, Karnik NS, Schueller SM, Zalta AK. Rates and correlates of well-being among youth experiencing homelessness. J Community Psychol. 2022 Sep;50(8):3746-3759. doi: 10.1002/jcop.22869. Epub 2022 Apr 23. PMID 35460583
- [Derived] Glover AC, Schueller SM, Winiarski DA, Smith DL, Karnik NS, Zalta AK. Automated Mobile Phone-Based Mental Health Resource for Homeless Youth: Pilot Study Assessing Feasibility and Acceptability. JMIR Ment Health. 2019 Oct 11;6(10):e15144. doi: 10.2196/15144. PMID 31605516

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT03776422/Prot_SAP_000.pdf